CLINICAL TRIAL: NCT03393923
Title: Effect of Anterior Wedge Use in Patients With Osteoarthritis Hip
Brief Title: Anterior Wedge in Patients With Osteoarthritis Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Claudio Cazarini Junior, Claudio Cazarini Júnior, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1112131232234
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2017-01

CONDITIONS: Gait, Frontal
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patient will undergo gait analysis
- Experimental group (Experimental): Patient will undergo gait analysis with use of anterior wedge
  Interventions: Other: Application of the anterior wedge

INTERVENTIONS:
Other: Application of the anterior wedge — Application of anterior wedge in tennis
  Arms: Experimental group

SUMMARY:
Ostearthritis is a great source of pain. In symptomatic hip the pain can lead the major disability and poor quality of life. Understand the musculoskeletal factores can lead to a better clinical management. The muscle strenghening of posterolateral complexo of hip is a important consideration. General Objective: Perform a Kinetic analysis 2D using na anterior wedge. Specific objective: Analyze the influence of posterolateral hip complex. Controlled clinical trial, composed by 30 individuals with and without osteoarthritis of hip e will be used a tools; Analogic Visual Scale, manual dynamometry to analyze force and kinetic analyze of gait through of Myovídeo analysis software.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary individuals
* Both genders
* Age equal to or greather than 50 years
* Diagnosis of osteoarthritis level II and III

Exclusion Criteria:

* fractures
* Neuromuscular diseases
* Other diseases of hip

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Inproved performance of the gluteus maximus | 24 hours
  Extent moment will be assessed by gait analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Flávia Nakatake, São Paulo, Brazil